CLINICAL TRIAL: NCT01493843
Title: A Phase II, Double-Blind, Placebo-Controlled, Randomized Study Evaluating the Safety and Efficacy of Carboplatin/Paclitaxel and Carboplatin/Paclitaxel/Bevacizumab With and Without GDC-0941 in Patients With Previously Untreated Advanced or Recurrent Non-small Cell Lung Cancer
Brief Title: Safety and Efficacy of Carboplatin/Paclitaxel and Carboplatin/Paclitaxel/Bevacizumab With and Without Pictilisib in Previously Untreated Advanced or Recurrent Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GO27912; 2011-002893-21 (EudraCT Number)
Record Dates: First submitted 2011-12-14; First posted 2011-12-16 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — 2-(1H-indazol-4-yl)-6-(4-methanesulfonylpiperazin-1-ylmethyl)-4-morpholin-4-ylthieno(3,2-d)pyrimidine; Bevacizumab; Carboplatin; Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Arm A: 340 mg pictilisib + CP (Experimental): Participants with advanced (Stage IV) or recurrent squamous NSCLC will be administered 340 mg pictilisib plus carboplatin (C) plus paclitaxel (P).
  Interventions: Drug: pictilisib; Drug: carboplatin; Drug: paclitaxel
- Arm B: Placebo + CP (Placebo Comparator): Participants with advanced (Stage IV) or recurrent squamous NSCLC will be administered placebo corresponding to 340 mg pictilisib plus carboplatin (C) plus paclitaxel (P). Participants with investigator assessed radiographic progression of NSCLC per RECIST 1.1 will be allowed to cross over to Arm A during the first 4 cycles with carboplatin + paclitaxel or after chemotherapy has been completed (Cycle >/= 5).
  Interventions: Drug: Placebo; Drug: carboplatin; Drug: paclitaxel
- Arm C: 340 mg pictilisib + CPB (Experimental): Participants with advanced (Stage IV) or recurrent non-squamous NSCLC will be administered 340 mg pictilisib plus carboplatin (C) plus paclitaxel (P) plus bevacizumab (B).
  Interventions: Drug: pictilisib; Drug: bevacizumab; Drug: carboplatin; Drug: paclitaxel
- Arm D: Placebo + CPB (Placebo Comparator): Participants with advanced (Stage IV) or recurrent non-squamous NSCLC will be administered placebo corresponding to 340 mg pictilisib plus carboplatin (C) plus paclitaxel (P). Participants with investigator assessed radiographic progression of NSCLC per RECIST 1.1 will be allowed to cross over to Arm C during the first 4 cycles with carboplatin + paclitaxel + bevacizumab or after chemotherapy has been completed (Cycle >/= 5).
  Interventions: Drug: Placebo; Drug: bevacizumab; Drug: carboplatin; Drug: paclitaxel
- Arm E: 260 mg pictilisib + CPB (Experimental): Participants with advanced (Stage IV) or recurrent non-squamous NSCLC will be administered 260 mg pictilisib plus carboplatin (C) plus paclitaxel (P) plus bevacizumab (B).
  Interventions: Drug: pictilisib; Drug: bevacizumab; Drug: carboplatin; Drug: paclitaxel
- Arm F: Placebo + CPB (Placebo Comparator): Participants with advanced (Stage IV) or recurrent non-squamous NSCLC will be administered placebo corresponding to 260 mg pictilisib plus carboplatin (C) plus paclitaxel (P). Participants with investigator assessed radiographic progression of NSCLC per RECIST 1.1 will be allowed to cross over to Arm E during the first 4 cycles with carboplatin + paclitaxel + bevacizumab or after chemotherapy has been completed (Cycle >/= 5).
  Interventions: Drug: Placebo; Drug: bevacizumab; Drug: carboplatin; Drug: paclitaxel

INTERVENTIONS:
Drug: pictilisib — Pictilisib, 260 milligrams (mg) or 340 mg, will be taken orally once daily on Days 1-14 of a 21-day cycle for four cycles. Starting with Cycle 5, pictilisib will be taken once daily continuously.
  Other Names: GDC-0941
  Arms: Arm A: 340 mg pictilisib + CP; Arm C: 340 mg pictilisib + CPB; Arm E: 260 mg pictilisib + CPB
Drug: Placebo — Placebo corresponding to 260 mg or 340 mg pictilisib will be taken orally once daily on Days 1-14 of a 21-day cycle for four cycles. Starting with Cycle 5, placebo will be taken once daily continuously.
  Arms: Arm B: Placebo + CP; Arm D: Placebo + CPB; Arm F: Placebo + CPB
Drug: bevacizumab — Bevacizumab, 15 milligrams per kilogram (mg/kg) will be administered intravenously (IV) at Day 1 of each 21-day cycle for a maximum of 34 cycles.
  Other Names: Avastin
  Arms: Arm C: 340 mg pictilisib + CPB; Arm D: Placebo + CPB; Arm E: 260 mg pictilisib + CPB; Arm F: Placebo + CPB
Drug: carboplatin — Carboplatin will be administered IV to achieve an initial target area under the concentration curve (AUC) of 6 milligrams per milliliter per minute (mg/mL per min) on Day 1 of each 21-day cycle for a maximum of four cycles.
Drug: paclitaxel — Paclitaxel will be administered at 200 milligrams per square meter (mg/m^2) IV on Day 1 of each 21-day cycle for a maximum of four cycles.

SUMMARY:
This multicenter, randomized, double-blind, placebo-controlled trial will evaluate the efficacy and safety of carboplatin/paclitaxel and carboplatin/paclitaxel/bevacizumab with and without pictilisib in particpants with previously untreated advanced or recurrent non-small cell lung cancer (NSCLC). Particpants will be randomized to receive 4 cycles of carboplatin (C)/paclitaxel (P) and either pictilisib or placebo, with (participants with non-squamous NSCLC) or without (participants with squamous NSCLC) bevacizumab (B). Anticipated time on study treatment is until disease progression or intolerable toxicity occurs. Participants in placebo arms with disease progression may cross over to open-label active pictilisib.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented advanced (Stage IV) or recurrent squamous (Arms A and B) or non-squamous (Arms C, D, E, and F) non-small cell lung cancer (NSCLC)
* Consent to the collection of an archival formalin-fixed paraffin-embedded (FFPE) block or freshly cut unstained tumor slides from archival tumor tissue or a newly collected tumor sample
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Disease that is measurable per Response Evaluation Criteria In Solid Tumors (RECIST) v1.1
* Adequate hematologic and end organ function
* Use of two effective forms of contraception

Exclusion Criteria:

* NSCLC with documented epidermal growth factor receptor (EGFR) mutation associated with response to EGFR inhibitors or documented fusion gene involving anaplastic lymphoma kinase (ALK) gene
* Prior therapy (including chemotherapy, antibody therapy, tyrosine kinase inhibitors, radiotherapy, immunotherapy, hormonal therapy, or investigational therapy) before Day 1 of Cycle 1 for the treatment of advanced (Stage IV) or recurrent NSCLC
* Known central nervous system (CNS) disease except for treated brain metastases
* Type I diabetes
* Type II diabetes requiring chronic therapy with insulin
* Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the participant at high risk for treatment complications
* Medical conditions that would contraindicate bevacizumab therapy in non-squamous NSCLC (Arms C, D, E, and F)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 501 (Actual)
Dates: Start 2012-01-20 (Actual); Primary Completion 2016-03-30 (Actual); Study Completion 2016-03-30 (Actual)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | Up to approximately 2.5 years
PFS in Participants with Phosphatidylinositol-4,5-Bisphosphate 3-Kinase Catalytic Subunit Alpha (PIK3CA) Amplification | Up to approximately 2.5 years
PFS in Participants with Phosphatase and Tensin Homolog (PTEN) Loss/Low | Up to approximately 2.5 years

SECONDARY OUTCOMES:
Objective Tumor Response | Up to approximately 2.5 years
Objective Tumor Response in Participants with PIK3CA Amplification | Up to approximately 2.5 years
Objective Tumor Response in Participants with PTEN Loss/low | Up to approximately 2.5 years
Duration of Objective Response (DoR) | Up to approximately 2.5 years
DoR in Participants with PIK3CA Amplification | Up to approximately 2.5 years
DoR in Participants with PTEN Loss/low | Up to approximately 2.5 years
Overall Survival (OS) | Up to approximately 2.5 years
OS in Participants with PIK3CA Amplification | Up to approximately 2.5 years
OS in Participants with PTEN Loss/low | Up to approximately 2.5 years
Percentage of Participants with Adverse Events | Up to approximately 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (120):
- United States (44):
  - Alabama Oncology, Birmingham, Alabama
  - Highlands Oncology Group, Rogers, Arkansas
  - cCare, Encinitas, California
  - Kaiser Permanente - Oakland, Oakland, California
  - Desert Hematology Oncology Group, Rancho Mirage, California
  - Kaiser Permanente - Roseville, Roseville, California
  - Kaiser Permanente Sacramento Medical Center, Sacramento, California
  - Southern CA Permanente Med Grp, San Diego, California
  - Kaiser Permanente, San Francisco, California
  - K. Permanente - Santa Clara, Santa Clara, California
  - Stockton Hema Onc Med Grp Inc, Stockton, California
  - Kaiser Permanente - Vallejo, Vallejo, California
  - K. Permanente - Walnut Creek, Walnut Creek, California
  - Hematology Oncology PC; Bennett Cancer Center, Stamford, Connecticut
  - Lynn Regional Cancer Center West, Boca Raton, Florida
  - Florida Cancer Specialists - Fort Myers (Colonial Center Dr), Fort Myers, Florida
  - Cancer Specialists; North Florida ;Jacksonville (AC Skinner Pkwy), Jacksonville, Florida
  - Advanced Medical Specialties, Miami, Florida
  - Florida Cancer Specialists (St. Petersburg - St. Anthony's Professional Building), St. Petersburg, Florida
  - University Cancer & Blood Center, LLC, Athens, Georgia
  - Peachtree Hematology & Oncology Consultants, Pc, Atlanta, Georgia
  - Georgia Cancer Specialists, Atlanta, Georgia
  - Hematology-Oncology of Indiana, Pc, Indianapolis, Indiana
  - Franklin Square Hospital, Baltimore, Maryland
  - Massachusetts General Hospital., Boston, Massachusetts
  - Dana Farber Cancer Inst., Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Wayne State University; Hemat/Onc, 4HW CRC, Detroit, Michigan
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Va Sierra Nevada Health Care System, Reno, Nevada
  - San Juan Oncology Associates, Farmington, New Mexico
  - Roswell Park Cancer Inst., Buffalo, New York
  - Piedmont Hematology Oncology Associates, Winston-Salem, North Carolina
  - Gabrail Cancer Center, Canton, Ohio
  - The Christ Hospital, Cincinnati, Ohio
  - Univ Hosp Case Medical Center, Cleveland, Ohio
  - Center for Biomedical Research LLC, Knoxville, Tennessee
  - The Sarah Cannon Research Inst, Nashville, Tennessee
  - Vanderbilt, Nashville, Tennessee
  - University of Texas M.D. Anderson Cancer Center, Houston, Texas
  - Wellmonth Physician Services, Bristol, Virginia
  - Blue Ridge Cancer Care - Roanoke, Roanoke, Virginia
  - VA Puget Sound Health Care Sys, Seattle, Washington
  - Northwest Medical Specialties, Tacoma, Washington
- Argentina (3):
  - Clinica Universitaria Reina Fabiola, Córdoba
  - Instituto FIDES, La Plata
  - Isis Centro Especializado de Luces; Oncology, Santa Fe
- Australia (7):
  - Royal Prince Alfred Hospital; Sydney Cancer Centre, Camperdown, New South Wales
  - St Vincent'S Hospital, Darlinghurst, New South Wales
  - Calvary Mater Newcastle; Medical Oncology, Waratah, New South Wales
  - Flinders Medical Centre; Medical Oncology, Bedford Park, South Australia
  - Royal Hobart Hospital; Medical Oncology, Hobart, Tasmania
  - Footscray Hospital, Footscray, Victoria
  - Royal Melbourne Hospital; Hematology and Medical Oncology, Parkville, Victoria
- Brazil (10):
  - Centro de Oncologia da Bahia - CENOB, Salvador, Estado de Bahia
  - Clinica de Tratamento e Pesquisa Oncologica - Oncotek, Brasília, Federal District
  - Instituto Nacional de Cancer - INCa; Oncologia, Rio de Janeiro, Rio de Janeiro
  - Liga Norte Riograndense Contra O Câncer, Natal, Rio Grande do Norte
  - Santa Casa de Misericordia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital Mae de Deus, Porto Alegre, Rio Grande do Sul
  - Centro de Pesquisas Oncologicas - CEPON, Florianópolis, Santa Catarina
  - Hospital Amaral Carvalho, Jaú, São Paulo
  - Instituto do Cancer do Estado de Sao Paulo - ICESP, São Paulo, São Paulo
  - Instituto de Oncologia de Sorocaba - CEPOS, Sorocaba, São Paulo
- Canada (2):
  - Mcgill University - Royal Victoria Hospital; Oncology, Montreal, Quebec
  - Hopital du Sacre-Coeur, Montreal, Quebec
- Chile (4):
  - Clinica Santa Maria, Santiago
  - Fundacion Arturo Lopez Perez, Santiago
  - Instituto Oncologico del sur, Temuco
  - Hospital Clinico Vina del Mar, Viña del Mar
- France (6):
  - Hopital Morvan, Brest
  - Clinique Victor Hugo; Radiotherapie, Le Mans
  - Clinique Catherine de Sienne; Service de cancérologie, Nantes
  - Ico Rene Gauducheau; Oncologie, Saint-Herblain
  - Centre Hospitalier de Villefranche sur Saone, Villefranche-sur-Saône
  - Institut Gustave Roussy; Departement Oncologie Medicale, Villejuif
- Germany (8):
  - Zentralklinik Bad Berka GmbH; Abteilung Onkologie und Hämatologie, Bad Berka
  - Asklepios-Fachkliniken Muenchen-Gauting; Onkologie, Gauting
  - Krankenhaus Grosshansdorf;Pneumologie & Thoraxchirurgie, Großhansdorf
  - St. Vincentius Kliniken Karlsruhe; Abteilung Hämatologie / Onkologie, Karlsruhe
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Medizinische Klinik, Pneumologie, Mainz
  - Universitätsklinikum Regensburg; Klinik und Poliklinik für Innere Medizin II, Pneumologie, Regensburg
  - Universitätsklinikum Ulm; Medizinische Uni-Klinik III Abt. Innere Medizin III Hämatologie u. Onkolo., Ulm
  - Schwarzwald-Baar Klinikum/VS GmbH; Onkologie/Hämatologie/Infektologie, Villingen-Schwenningen
- Hungary (6):
  - Orszagos Koranyi TBC es Pulmonologiai Intezet, Budapest
  - Koch Robert Korhaz, Edelény
  - Veszprem Megyei Onkormanyzat Tudogyogyintezet, Farkasgyepű
  - Vas Megyei Markusovszky Korhaz ; Pulmonology, Szombathely
  - Tudogyogyintezet Torokbalint, Törökbálint
  - Zala Megyei Korhaz; Dept of Pulmonary Medicine, Zalaegerszeg
- Israel (3):
  - Shaare Zedek Medical Center; Oncology Dept, Jerusalem
  - Meir Medical Center; Oncology, Kfar Saba
  - Chaim Sheba Medical Center; Oncology Dept, Ramat Gan
- Italy (5):
  - Ausl Di Bologna-Ospedale Bellaria;U.O. Oncologia Medica, Bologna, Emilia-Romagna
  - Irccs Centro Di Riferimento Oncologico (CRO); Dipartimento Di Oncologia Medica, Aviano, Friuli Venezia Giulia
  - ASST DI MONZA; Oncologia Medica, Monza, Lombardy
  - Az. Osp. S. Luigi Gonzaga; Malattie Apparato Respiratorio 5 Ad Indirizzo Oncologico, Orbassano, Piedmont
  - A.O.U.I. VERONA-OSPEDALE POLICLINICO G.B. ROSSI BORGO ROMA;ONCOLOGIA MEDICA-d.U., Verona, Veneto
- Netherlands (3):
  - Amphia Ziekenhuis, Breda
  - Catharina-ziekenhuis; Longgeneeskunde en Tuberculose, Eindhoven
  - Universitair Medisch Centrum Groningen, Groningen
- Russia (5):
  - Regional Oncology Center, Chelyabinsk
  - Moscow city oncology hospital #62 of Moscow Healthcare Department, Moscow
  - City Oncology Hospital; Chemotherapy Dept, Nizhny Novgorod
  - Rsrch Onc Inst of Rosmed Tech; n.a. prof. N.N. Petrov; Dept of Surgery, Saint Petersburg
  - Leningrad Regional Clinical Hospital, Saint Petersburg
- Spain (5):
  - Hospital Nuestra Señora de Sonsoles; servicio de Oncologia, Ávila
  - Hospital Univ Vall d'Hebron; Servicio de Oncologia, Barcelona
  - Hospital Universitari Germans Trias i Pujol; Servicio de Oncologia, Barcelona
  - Hospital Universitario 12 de Octubre; Servicio de Oncologia, Madrid
  - Hospital Universitario Puerta de Hierro; Servicio de Oncologia, Madrid
- Ukraine (6):
  - Kiev City Clinical Oncology Center, Kiev
  - Volyn Regional Oncology Dispensary, Lutsk
  - State Oncology Regional Treatment-Diagnostic Center; Chemotherapy Department, Lviv
  - Crimean Republican Institute; Oncology Clin Dispensary; Chemotherapy Dept, Simferopol
  - Sumy Reg. Clin. Oncological Dispensary; Thoracall Department, Sumy
  - Zaporizhzhia Regional Clinical Oncology Dispensary; Zaporizhzhya State Medical University, Zaporizhzhya
- United Kingdom (3):
  - Royal Surrey County Hospital; St. Lukes Cancer Centre, Guildford
  - Leicester Royal Infirmary; Dept. of Medical Oncology, Leicester
  - Christie Hospital Nhs Trust; Medical Oncology, Manchester